CLINICAL TRIAL: NCT05229692
Title: Effect of Neuromuscular Electrical Stimulation on the Post-Operative Abdominoplasty Patient.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of interest from participants
Sponsor: NeuFit - Neurological Fitness and Education (Industry)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000863
Record Dates: First submitted 2021-08-23; First posted 2022-02-08 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Rectus Diastasis
Keywords: abdominoplasty; NEUBIE; neuromuscular electrical stimulation; rectus diastatis

STUDY DESIGN:
Intervention Model Description: Study will be divided into two randomly assigned groups - control and interventional. Control group will receive current standard of care for recovery (rest and minimal activity for 6 weeks post-operative). Interventional group will receive neuromuscular electrical stimulation treatments 2 times a week for 6 weeks post-operative.
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed at Piazza Surgical Center. Assessors will be blinded to which intervention participant has received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NEUBIE (Experimental): Experimental group will receive rehabilitation training with the NEUBIE for 6 weeks post-operative. Training will occur at Neufit 2x a week from week 1-5, and will be administered by NeuFit clinic staff. Exercises and ability to complete exercises will be recorded by NeuFit staff in standardized clinic evaluation forms.
  Participants will undergo will undergo both active muscle tests and body analysis tests.
  Measurements will be taken at The Piazza Center by clinic staff prior to surgery at 2,4,6,8, and 12 weeks post-operative. Measurements will be used to demonstrate milestones of functional recovery, comparable between subjects by weeks achieved.
  Interventions: Device: NEUBIE
- Control (No Intervention): Control group will receive current post-operative standard of care for abdominoplasty, which includes using an abdominal binder, rest and minimal activity for 6 weeks.
  Participants will undergo both active muscle tests and body analysis tests. Measurements will be taken at The Piazza Center by clinic staff prior to surgery at 2,4,6,8, and 12 weeks post-operative. Measurements will be used to demonstrate milestones of functional recovery, comparable between subjects by weeks achieved.

INTERVENTIONS:
Device: NEUBIE — Participants will be asked to undergo electrical stimulation with the NEUBIE at their "treatment threshold". Treatment threshold will be described as "uncomfortable," but not "painful" (a 7 out of 10 on a perceived intensity scale).
  Session length: ≤ 30 minutes Treatment frequency: 2x per week for 5 weeks
  Week 1 post-op (treatments 1-2) Activity: Passive Neubie on Abdominals & Obliques
  Weeks 2-3 (treatments 3-6)
  * Passive Neubie
  * Isometric movements with Neubie on abdominals and obliques
  * Active mobilizations with Neubie on abdominals and obliques
  Weeks 4-5 (treatments 7-10)
  * Active mobilizations with Neubie on abdominals and obliques
  * Core Strength Exercise circuit with Neubie on abdominals and obliques
  Other Names: NeuFit
  Arms: NEUBIE

SUMMARY:
The purpose of this study is to determine the impact of rehabilitative training of the abdominal wall with direct current neuromuscular electrical stimulation (the NEUBIE device) on recovery time from abdominoplasty (tummy tuck).

DETAILED DESCRIPTION:
Participants will undergo abdominoplasty surgery and begin rehabilitation training within the first week post-operation. Standardized measurements of recovery progress will be taken starting prior to operation, and at 2, 4, 6, 8 and 12 weeks post-operation. Participants will undergo either the traditional standard of care of rest, with minimal activity for at least 6 weeks (control group) or a 5 week training course with the NEUBIE (experimental group), starting with passive electrical stimulation in the first week post-operation, and moving towards more advanced abdominal movements accompanied with stimulation in the subsequent four weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Rectus Diastasis
2. Previous pregnancy
3. Excess localized adiposity in the lower abdomen
4. Excess atrophic skin of the abdomen
5. Physician clearance to participate
6. Scheduled for full abdominoplasty (no mini-abdominoplasty included)

Exclusion Criteria:

1. Currently pregnant
2. Cardiac Pacemaker
3. Active or recent cancer in the abdominal area
4. Active or recent blood clots in the abdominal area
5. History of epilepsy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Bio-impedance analysis muscle mass | Pre-intervention
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure muscle mass.
Bio-impedance analysis trunk fat | Pre-intervention
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure body fat.
Bio-impedance analysis trunk mass | Pre-intervention
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk mass.
Bio-impedance analysis muscle mass | 2 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure muscle mass.
Bio-impedance analysis trunk fat | 2 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk body fat.
Bio-impedance analysis trunk mass | 2 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk mass.
Bio-impedance analysis muscle mass | 4 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure muscle mass.
Bio-impedance analysis trunk fat | 4 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk body fat.
Bio-impedance analysis trunk mass | 4 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk mass.
Bio-impedance analysis muscle mass | 6 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure muscle mass.
Bio-impedance analysis trunk fat | 6 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk body fat.
Bio-impedance analysis trunk mass | 6 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk mass.
Bio-impedance analysis muscle mass | 8 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure muscle mass.
Bio-impedance analysis trunk fat | 8 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk body fat.
Bio-impedance analysis trunk mass | 8 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk mass.
Bio-impedance analysis muscle mass | 12 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure muscle mass.
Bio-impedance analysis trunk fat | 12 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk body fat.
Bio-impedance analysis muscle mass | 12 weeks
  Bioelectrical impedance analysis is a method for estimating body composition, in particular body fat and muscle mass, where a weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body. Here it will be used to measure trunk mass.
Range of Motion | Pre-intervention
  Range of motion is determined via a goniometer. Body is moved in specific directions and goniometer is used to measure the amount of motion that occurs.
Range of Motion | 2 weeks
  Range of motion is determined via a goniometer. Body is moved in specific directions and goniometer is used to measure the amount of motion that occurs.
Range of Motion | 4 weeks
  Range of motion is determined via a goniometer. Body is moved in specific directions and goniometer is used to measure the amount of motion that occurs.
Range of Motion | 6 weeks
  Range of motion is determined via a goniometer. Body is moved in specific directions and goniometer is used to measure the amount of motion that occurs.
Range of Motion | 8 weeks
  Range of motion is determined via a goniometer. Body is moved in specific directions and goniometer is used to measure the amount of motion that occurs.
Range of Motion | 12 weeks
  Range of motion is determined via a goniometer. Body is moved in specific directions and goniometer is used to measure the amount of motion that occurs.
Core strength and endurance bridge | Pre-intervention
  Core strength and endurance will be measured by duration of ability to hold a glute bridge.
Core strength and endurance plank | Pre-intervention
  Core strength and endurance will be measured by duration of ability to hold a plank.
Core strength and endurance bridge | 2 weeks
  Core strength and endurance will be measured by duration of ability to hold a glute bridge.
Core strength and endurance plank | 2 weeks
  Core strength and endurance will be measured by duration of ability to hold a glute bridge.
Core strength and endurance plank | 4 weeks
  Core strength and endurance will be measured by duration of ability to hold a plank.
Core strength and endurance bridge | 4 weeks
  Core strength and endurance will be measured by duration of ability to hold a glute bridge.
Core strength and endurance plank | 6 weeks
  Core strength and endurance will be measured by duration of ability to hold a plank.
Core strength and endurance bridge | 6 weeks
  Core strength and endurance will be measured by duration of ability to hold a glute bridge.
Core strength and endurance plank | 8 weeks
  Core strength and endurance will be measured by duration of ability to hold a plank.
Core strength and endurance bridge | 8 weeks
  Core strength and endurance will be measured by duration of ability to hold a glute bridge.
Core strength and endurance plank | 12 weeks
  Core strength and endurance will be measured by duration of ability to hold a plank.
Core strength and endurance bridge | 12 weeks
  Core strength and endurance will be measured by duration of ability to hold a glute bridge.
Lower abdominal strength | Pre-intervention
  Lower abdominal strength will be measured by ability to perform an eccentric double leg lowering movement.
Lower abdominal strength | 2 weeks
  Lower abdominal strength will be measured by ability to perform an eccentric double leg lowering movement.
Lower abdominal strength | 4 weeks
  Lower abdominal strength will be measured by ability to perform an eccentric double leg lowering movement.
Lower abdominal strength | 6 weeks
  Lower abdominal strength will be measured by ability to perform an eccentric double leg lowering movement.
Lower abdominal strength | 8 weeks
  Lower abdominal strength will be measured by ability to perform an eccentric double leg lowering movement.
Lower abdominal strength | 12 weeks
  Lower abdominal strength will be measured by ability to perform an eccentric double leg lowering movement.
Sit up Test | Pre-intervention
  Ability to complete a sit up will be measured as a general measurement of core strength and range of motion.
Sit up Test | 2 weeks
  Ability to complete a sit up will be measured as a general measurement of core strength and range of motion.
Sit up Test | 4 weeks
  Ability to complete a sit up will be measured as a general measurement of core strength and range of motion.
Sit up Test | 6 weeks
  Ability to complete a sit up will be measured as a general measurement of core strength and range of motion.
Sit up Test | 8 weeks
  Ability to complete a sit up will be measured as a general measurement of core strength and range of motion.
Sit up Test | 12 weeks
  Ability to complete a sit up will be measured as a general measurement of core strength and range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Piazza, MD, Principal Investigator — University of Texas at Austin
Locations (1):
- Piazza Center for Plastic Surgery and Advanced Skin Care, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thakral G, Lafontaine J, Najafi B, Talal TK, Kim P, Lavery LA. Electrical stimulation to accelerate wound healing. Diabet Foot Ankle. 2013 Sep 16;4. doi: 10.3402/dfa.v4i0.22081. PMID 24049559
- [Background] Ud-Din S, Bayat A. Electrical Stimulation and Cutaneous Wound Healing: A Review of Clinical Evidence. Healthcare (Basel). 2014 Oct 27;2(4):445-67. doi: 10.3390/healthcare2040445. PMID 27429287
- [Background] da Silva MP, Liebano RE, Rodrigues VA, Abla LE, Ferreira LM. Transcutaneous electrical nerve stimulation for pain relief after liposuction: a randomized controlled trial. Aesthetic Plast Surg. 2015 Apr;39(2):262-9. doi: 10.1007/s00266-015-0451-6. Epub 2015 Feb 10. PMID 25665520
- [Background] Klika AK, Yakubek G, Piuzzi N, Calabrese G, Barsoum WK, Higuera CA. Neuromuscular Electrical Stimulation Use after Total Knee Arthroplasty Improves Early Return to Function: A Randomized Trial. J Knee Surg. 2022 Jan;35(1):104-111. doi: 10.1055/s-0040-1713420. Epub 2020 Jul 1. PMID 32610358
- [Background] Delanois R, Sodhi N, Acuna A, Doll K, Mont MA, Bhave A. Use of home neuromuscular electrical stimulation in the first 6 weeks improves function and reduces pain after primary total knee arthroplasty: a matched comparison. Ann Transl Med. 2019 Oct;7(Suppl 7):S254. doi: 10.21037/atm.2019.09.150. PMID 31728378
- [Background] Demircioglu DT, Paker N, Erbil E, Bugdayci D, Emre TY. The effect of neuromuscular electrical stimulation on functional status and quality of life after knee arthroplasty: a randomized controlled study. J Phys Ther Sci. 2015 Aug;27(8):2501-6. doi: 10.1589/jpts.27.2501. Epub 2015 Aug 21. PMID 26355656
- [Background] Bistolfi A, Zanovello J, Ferracini R, Allisiardi F, Lioce E, Magistroni E, Berchialla P, Da Rold I, Massazza G. Evaluation of the Effectiveness of Neuromuscular Electrical Stimulation After Total Knee Arthroplasty: A Meta-Analysis. Am J Phys Med Rehabil. 2018 Feb;97(2):123-130. doi: 10.1097/PHM.0000000000000847. PMID 29016401
- [Background] Yue C, Zhang X, Zhu Y, Jia Y, Wang H, Liu Y. Systematic Review of Three Electrical Stimulation Techniques for Rehabilitation After Total Knee Arthroplasty. J Arthroplasty. 2018 Jul;33(7):2330-2337. doi: 10.1016/j.arth.2018.01.070. Epub 2018 Feb 6. PMID 29530519